CLINICAL TRIAL: NCT03454464
Title: To Evaluate the Practicable, Thoroughness and Clinical Value of Bilateral Central Compartment Dissection While Preserve Contrary Thyroid Glands
Brief Title: Evaluation of Central Compartment Dissection Without Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Clinical professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD
Record Dates: First submitted 2018-02-07; First posted 2018-03-06 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Thyroidectomy; Thyroid Cancer; Central Compartment Neck Dissction
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional operation group (Sham Comparator): Conventional operation group,Thyroidectomy was performed first, and central compartment dissection was performed. This is a routine procedure.
  Interventions: Procedure: Conventional
- central neck dissection first group (Experimental): central neck dissection first group,after FNA confirmed of thyroid carcinoma, the central compartment neck dissection was carried out before thyroidectomy , finally complement of central compartment neck dissection.
  Interventions: Procedure: central neck dissection first

INTERVENTIONS:
Procedure: Conventional — Conventional operation ,Thyroidectomy was performed first, and central compartment dissection was performed. This is a routine procedure
  Arms: Conventional operation group
Procedure: central neck dissection first — central neck dissection first ,after FNA confirmed of thyroid carcinoma, the central compartment neck dissection was carried out before thyroidectomy , finally complement of central compartment neck dissection.
  Arms: central neck dissection first group

SUMMARY:
In accordance with the current guidelines,papillary thyroid microcarcinoma such as turmo invasive nerve or trachea, requires total thyroidectomy for follow-up iodine-131 treatment.In the course of clinical work, if the patient can achieve R0 resection, most of the patients do not need iodine-131 treatment,Therefore, there is no need to continue total thyroidectomy.To evaluate the practicable, thoroughness and Clinical value of bilateral central compartment dissection while preserve contrary thyroid glands.

DETAILED DESCRIPTION:
In accordance with the current guidelines,papillary thyroid microcarcinoma such as turmo invasive nerve or trachea, requires total thyroidectomy for follow-up iodine-131 treatment.In the course of clinical work, if the patient can achieve R0 resection, most of the patients do not need iodine-131 treatment,Therefore, there is no need to continue total thyroidectomy.This study assesses new procedures by adjusting the sequence of procedures. complications and the thoroughness of the operation were evaluated, thus Clinical value of bilateral central compartment dissection with preserve contrary thyroid glands were ananlyed.

ELIGIBILITY:
Inclusion Criteria:

Tumor diameter less than 1cm The tumor is located in the lower part of the gland No lateral cervical lymph node metastases Traditional open surgery

Exclusion Criteria:

Select the endoscopic surgery or robotic surgery patients Tumor invades the surrounding trachea and esophagus Patients refused to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
number of the lymph node | 2 day post operation
  the number of the lymph node
number of postive lymph node | 2 day post operation
  The number of postive lymph node
The weight of the central compartment tissue. | introoperation
  The weight of the central compartment tissue.

SECONDARY OUTCOMES:
thyroid volume | The day before the operation
  thyroid volume
recurrent laryngeal nerve palsy | 1 day ,2weeks,3months,6months post operation
  the number of recurrent laryngeal nerve palsy

CONTACTS AND LOCATIONS:
Overall Officials: wen-xin zhao, md, Study Director — fujian meidcal university
Locations (1):
- Wen-xin ZHAO, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided